CLINICAL TRIAL: NCT01855919
Title: Effect of Duloxetine 60 mg Versus Placebo in Patients With Chronic Low Back Pain in Japan
Brief Title: A Study of Duloxetine (LY248686) in Participants With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14376; F1J-JE-HMGY (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Chronic Low Back Pain; CLBP
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine 20 milligram (mg) for first week, 40 mg for second week and 60 mg for next 12 weeks administered orally once daily. Tapering week doses of 40 mg for first 3 days and 20 mg for last 4 days of week.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo administered orally once every day for 15 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy and safety of duloxetine in participants with Chronic Low Back Pain (CLBP).

ELIGIBILITY:
Inclusion Criteria:

* Participants with CLBP present for the preceding 6 months or longer
* Participants used nonsteroidal anti-inflammatory drugs for CLBP for more than 14 days on average per month in the past 3 months and more than 14 days in one month prior to screening
* Participants having a score of ≥4 on Brief Pain Inventory (BPI) average pain score before randomized
* Female participants having child-bearing potential must test negative (-) on a pregnancy test

Exclusion Criteria:

* Participants have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication
* Participants having a history of low back surgery
* Participants having received epidural steroids, facet block, nerve block or other invasive procedures aimed to reduce low back pain within one month prior to screening
* Participants who have any difficulties to fulfill diary appropriately
* Participants having any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder
* Participants having major depressive disorder as determined using depression module of the Mini-International Neuropsychiatric Interview
* Participants having primary painful condition due to other than CLBP
* Participants being anticipated by the investigator to require use of nonsteroidal anti-inflammatory drugs and includes acetaminophen, opioid analgesics, or other excluded medication for the duration of the study
* Participants being considered as inappropriate for participation to the study for any medical or other reason as judged by the investigator
* Participants answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring within the past month (Columbia Suicide Severity Rating Scale, Suicide Ideation section - Questions 4 and 5; Suicidal Behavior section)
* Participants having a positive urine drug screen for any substances of abuse or excluded medication
* Participants having alanine aminotransferase or aspartate aminotransferase higher than 100 International Units per Liter (IU/L) or total bilirubin higher than 1.6 milligram per deciliter (mg/dL)
* Participants having serum creatinine level higher than 2.0 mg/dL, or had renal transplantation or receiving renal dialysis
* Participants having uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension
* Participants have had previous exposure to duloxetine or completed / withdrawn from any study investigating duloxetine
* Participants having serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions that, in the opinion of investigator, would compromise participation or be likely to lead to hospitalization during the course of the study
* Participants have known hypersensitivity to multiple medications
* Participants having diagnosis seronegative spondyloarthropathy or rheumatoid arthritis
* Participants taking any excluded medications that cannot be discontinued
* Participants treating with a monoamine oxidase inhibitor (MAOI) within 14 days or the potential need to use an MAOI during the study or within 5 days of discontinuation of study drug
* Participants are non-ambulatory or require the use of crutches or a walker
* Participants having a history of substance abuse or dependence within the past year, excluding nicotine and caffeine
* Pregnant participants or participants were breast-feeding, or wished to be pregnant during the clinical trial period
* Participants cannot use appropriate contraceptive method or do not want to use that from screening until one month after the end of administration of the investigational drug

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama, Japan

REFERENCES:
- [Derived] Enomoto H, Sasaki N, Fujikoshi S, Yoshikawa A, Tsuji T, Takeshita K. Relationship Between Pain Alleviation and Disease-specific Health-related Quality of Life Measures in Patients With Chronic Low Back Pain Receiving Duloxetine: Exploratory Post Hoc Analysis of a Japanese Phase 3 Randomized Study. J Am Acad Orthop Surg Glob Res Rev. 2019 Nov 27;3(11):e18.00086. doi: 10.5435/JAAOSGlobal-D-18-00086. eCollection 2019 Nov. PMID 31875196
- [Derived] Tsuji T, Itoh N, Ishida M, Ochiai T, Konno S. Response to duloxetine in chronic low back pain: exploratory post hoc analysis of a Japanese Phase III randomized study. J Pain Res. 2017 Sep 4;10:2157-2168. doi: 10.2147/JPR.S138172. eCollection 2017. PMID 28919811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow includes information on participants who completed the study. 2 participants who were assigned to receive placebo received duloxetine instead. These participants were treated as placebo in efficacy analysis and as duloxetine in safety analysis. In the participant flow, these participants are included under placebo.
Groups:
- Duloxetine: Duloxetine 20 milligram (mg) during Week 1, 40 mg during Week 2, and 60 mg during Weeks 3 to 14 administered in capsule form orally once daily. Tapering doses of 40 mg for first 3 days and 20 mg for last 4 days were administered during Week 15.
- Placebo: Placebo administered in capsule form orally once every day for 15 weeks.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 232 | 226
Received at Least 1 Dose of Study Drug | 232 | 226
Completed | 209 | 200
Not Completed | 23 | 26
Not completed — Adverse Event | 16 | 8
Not completed — Lack of Efficacy | 1 | 3
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Protocol Violation | 1 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose Brief Pain Inventory (BPI) pain severity (average pain) scores.
Groups:
- Duloxetine: Duloxetine 20 mg during Week 1, 40 mg during Week 2, and 60 mg during Weeks 3 to 14 administered in capsule form orally once daily. Tapering doses of 40 mg for first 3 days and 20 mg for last 4 days were administered during Week 15.
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 230 | 226 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (13.2) | 57.8 (13.7) | 58.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 122 | 237
  Male | 115 | 104 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 230 | 226 | 456
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 230 | 226 | 456
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 230 | 226 | 456

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 14 in Brief Pain Inventory (BPI) 24-Hour Average Pain Severity Item
Description: BPI is a self-reported scale that measures the severity of pain based on the average pain during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). Higher scores indicated worsening of pain. Least squares (LS) means calculated using mixed model repeating measure (MMRM) adjusted for treatment, visit, interaction between treatment and visit as fixed effects and baseline value as covariate.
Time Frame: Baseline, Week 14
Population: FAS: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) scores.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | -2.43 (0.11) | -1.96 (0.11)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.77 to -0.16]

2. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at Week 14
Description: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse). LS means calculated using MMRM adjusted for treatment, visit, interaction between treatment and visit as fixed effects and baseline value as covariate.
Time Frame: Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | 2.46 (0.07) | 2.76 (0.07)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.48 to -0.10]

3. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ-24) to Week 14
Description: The RMDQ-24 is a health status measure completed by participants to assess physical disability due to low back pain. Participants answered 24 questions about impairment of daily living activities (standing, walking, sitting, wearing clothes, working, etc.) resulting from low back pain. The number of statements marked was summed by the clinician for a total score. The total scores range from 0 (no disability) to 24 (severe disability). LS means calculated using analysis of covariance (ANCOVA) with treatment group as a fixed effect, and baseline value as a covariate.
Time Frame: Baseline, Week 14
Population: FAS: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) scores. The last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | -3.86 (0.22) | -3.23 (0.22)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0439, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.25 to -0.02]

4. Secondary Outcome: Change From Baseline in BPI Pain Severity Items (BPI-S) and Interference Items (BPI-I) Scores to Week 14
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores range from: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores range from: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference is defined as the average of non-missing scores of individual interference items. Higher scores indicated worsening of pain. LS means calculated using MMRM adjusted for treatment, visit, interaction between treatment and visit as fixed effects and baseline value as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale
  Worst Pain | -2.63 (0.13) | -2.33 (0.13)
  Least Pain | -1.69 (0.10) | -1.19 (0.11)
  Current Pain | -2.42 (0.12) | -2.03 (0.12)
  General Activity | -2.46 (0.13) | -2.16 (0.13)
  Mood | -2.15 (0.11) | -1.83 (0.11)
  Walking Ability | -2.05 (0.11) | -1.92 (0.11)
  Normal Work | -2.17 (0.12) | -2.17 (0.12)
  Relationship People | -1.02 (0.10) | -0.98 (0.10)
  Sleep | -1.41 (0.11) | -1.40 (0.11)
  Enjoyment of Life | -1.52 (0.11) | -1.48 (0.11)
  Average of 7 Interference Items | -1.83 (0.10) | -1.70 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.1010, Mixed Models Analysis — p-value is for worst pain; Median Difference (Final Values) = -0.30, 95% CI 2-sided [-0.66 to 0.06]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — p-value is for least pain; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.79 to -0.21]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0230, Mixed Models Analysis — p-value is for Pain Right Now; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.74 to -0.05]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0874, Mixed Models Analysis — p-value is for General Activity; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.66 to 0.05]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0436, Mixed Models Analysis — p-value is for Mood; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.63 to -0.01]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.3902, Mixed Models Analysis — p-value is for Walking Ability; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.45 to 0.18]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.9910, Mixed Models Analysis — p-value is for Normal Work; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.33 to 0.33]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.7848, Mixed Models Analysis — p-value is for Relationship People; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.30 to 0.23]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.9424, Mixed Models Analysis — p-value is for Sleep; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.32 to 0.30]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.7932, Mixed Models Analysis — p-value is for Enjoyment of Life; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.35 to 0.27]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.3761, Mixed Models Analysis — p-value is for Average of 7 Items; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.40 to 0.15]

5. Secondary Outcome: Change From Baseline in Weekly Mean of 24 Hour Average Pain and Worst Daily Pain Severity Scores to Week 14
Description: 24-hour average pain severity scores were recorded daily on an 11-point Likert scale, an ordinal scale, with scores ranging from 0 (no pain) to 10 (worst possible pain). The 11-point Likert scale was also used for assessment of average pain and worst pain within 24-hours. For the analysis, weekly mean was calculated. LS means calculated using MMRM adjusted for treatment, week, interaction between treatment and week as fixed effects and baseline value as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale
  Average Pain | -2.15 (0.10) | -1.73 (0.11)
  Worst Pain | -2.25 (0.12) | -1.91 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis — p-value is for Average Pain; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.71 to -0.13]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0442, Mixed Models Analysis — p-value is for Worst pain; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.69 to -0.01]

6. Secondary Outcome: Percentage of Participants With Reduction of ≥30% and ≥50% in BPI Average Pain Score at Week 14
Description: Pain severity was measured using an 11 point BPI scale from 0 (no pain) to 10 (worst pain) to determine average pain in the past 24 hours (average pain). A 30% (or 50%) improvement was defined as a ≥30% (or ≥50%) reduction in BPI pain severity from baseline to endpoint. Percentage of participants = (number of participants with ≥30% or ≥50% pain reduction / total number of participants in treatment group) * 100.
Time Frame: Baseline, Week 14
Population: FAS: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) scores. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
percentage of participants
  ≥30% pain reduction | 68.7 | 52.2
  ≥50% pain reduction | 56.5 | 39.4
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0003, Mantel Haenszel — p-value is for ≥30%; Risk Ratio (RR) = 1.31, 95% CI 2-sided [1.13 to 1.53]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0003, Mantel Haenszel — p-value is for ≥50%; Risk Ratio (RR) = 1.43, 95% CI 2-sided [1.18 to 1.75]

7. Secondary Outcome: Percentage of Participants With Sustained Pain Reduction in BPI Average Pain Score
Description: Pain severity was measured using an 11 point BPI scale from 0 (no pain) to 10(worst pain) to determine average pain in the past 24 hours (average pain). Participants were considered to have sustained pain reduction of ≥30% in the BPI-severity score (average pain) at the time of final evaluation and at least 1 other time point prior to the time of final evaluation compared with baseline, and a reduction of ≥20% from baseline sustained at all evaluation time points between that period. Percentage of participants = (number of participants with sustained pain reduction / total number of participants in treatment group) * 100.
Time Frame: Baseline through Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
percentage of participants | 61.3 | 46.0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0012, Mantel Haenszel; Risk Ratio (RR) = 1.33, 95% CI 2-sided [1.12 to 1.58]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-Severity) to Week 14
Description: CSI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). LS means calculated using MMRM adjusted for treatment, visit, interaction between treatment and visit as fixed effects and baseline value as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | -1.46 (0.06) | -1.17 (0.06)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.46 to -0.10]

9. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) to Week 14
Description: BDI-II is a 21-question multiple-choice self-reported inventory about depressive symptoms (sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping patterns, irritability, changes in appetite, concentration difficulties, tiredness or fatigue, and loss of interest in sex). The scores for each item range from 0 (best) to 3 (worst) with possible total scores of 0 to 63, where higher total scores indicate more severe depressive symptoms. LS means calculated using ANCOVA adjusted for treatment, as fixed effect and baseline as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | -1.39 (0.24) | -1.04 (0.24)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.3012, ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.03 to 0.32]

10. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) to Week 14
Description: SF-36 Health Status Survey is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. LS means calculated using ANCOVA adjusted for treatment, as fixed effect and baseline as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: Duloxetine 20 milligram (mg) for first week, 40 mg for second week and 60 mg for next 12 weeks administered in capsule form orally once daily. Tapering doses of 40 mg for first 3 days and 20 mg for last 4 days were administered during the last week.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale
  Physical Functioning | 8.47 (0.79) | 7.20 (0.80)
  Role (Physical) | 10.58 (1.15) | 10.00 (1.16)
  Bodily Pain | 12.56 (0.94) | 11.01 (0.95)
  General Health | 6.72 (0.85) | 3.78 (0.86)
  Vitality | 5.56 (0.97) | 4.41 (0.97)
  Social Functioning | 6.40 (1.00) | 4.77 (1.01)
  Role (Emotional) | 5.78 (1.13) | 6.18 (1.14)
  Mental Health | 5.63 (0.81) | 2.42 (0.82)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.2581, ANCOVA — p-value for Physical Functioning; Mean Difference (Final Values) = 1.27, 95% CI 2-sided [-0.93 to 3.47]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.7208, ANCOVA — p-value for Role (Physical); Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-2.62 to 3.79]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.2487, ANCOVA — p-value for Bodily Pain; Mean Difference (Final Values) = 1.55, 95% CI 2-sided [-1.09 to 4.19]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0151, ANCOVA — p-value for General Health; Mean Difference (Final Values) = 2.94, 95% CI 2-sided [0.57 to 5.31]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.4000, ANCOVA — p-value for Vitality; Mean Difference (Final Values) = 1.16, 95% CI 2-sided [-1.54 to 3.85]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.2529, ANCOVA — p-value for Social Functioning; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [-1.17 to 4.43]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.8042, ANCOVA — p-value for Role(Emotional); Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-3.55 to 2.75]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0058, ANCOVA — p-value is for Mental Health; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [0.94 to 5.48]

11. Secondary Outcome: Change From Baseline in European Quality of Life Questionnaire-5 Dimension (EQ-5D) to Week 14
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3 level scale (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm ranging from -0.111 to 1.0, with higher scores indicating better quality of life. LS means calculated using ANCOVA adjusted for treatment, as fixed effect and baseline as covariate.
Time Frame: Baseline, Week 14
Population: FAS: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-dose BPI pain severity (average pain) scores. LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
units on a scale | 0.09 (0.01) | 0.08 (0.01)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.5237, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.02 to 0.03]

12. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Instrument to Week 14
Description: WPAI is a self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities, and yields 4 types of scores: Absenteeism (work time missed)=Question (Q)2/(Q2+4))*100); Presenteeism (impairment at work/reduced on-the-job effectiveness)=(Q5/10)*100); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism)=(Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)])*100); and Activity Impairment=(Q6/10)*100. Scores range from 0 to 1 for each of the above 4 types; higher scores indicate greater impairment. LS means calculated using ANCOVA adjusted for treatment, as fixed effect and baseline as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 230 | 226
hours
  Work time missed (n=135, 140) | -0.01 (0.01) | 0.02 (0.01)
  Impairment at work (n=136, 140) | -0.13 (0.02) | -0.09 (0.02)
  Work productivity loss (n=135, 140) | -0.13 (0.02) | -0.09 (0.02)
  Work activity impairment (n=230, 226) | -0.14 (0.01) | -0.12 (0.01)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0460, ANCOVA — p-value for Work time missed; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.00]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0753, ANCOVA — p-value for Impairment at work; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.08 to 0.00]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.0795, ANCOVA — p-value for Work productivity loss; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.08 to 0.00]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.1466, ANCOVA — p-value for Work activity impairment; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.06 to 0.01]

13. Secondary Outcome: Number of Participants With Suicidal Thoughts And Behaviors During Study [Columbia Suicide Severity Rating Scale (C-SSRS)]
Description: C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any 1 of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any 1 of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline through Week 14
Population: All randomized participants who received at least 1 dose of study drug, responded no at baseline to the suicide related questionnaire and had data at post-treatment for each question.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 232 | 224
percentage of participants
  Wish to be dead (n=226, 220) | 0 | 0
  Nonspecific active suicidal thoughts (n=231, 223) | 0 | 0
  Suicidal behavior (n=232, 224) | 0 | 0

14. Secondary Outcome: Percentage of Participants With Fall Events in Fall Questionnaire
Description: Participants evaluated their experience with and details of falls which were recorded. Percentage = (number of participants with fall events) /(total in treatment group) * 100.
Time Frame: Baseline through Week 14
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 234 | 224
percentage of participants | 10.3 | 8.0

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 4/234 | 4/224
Other Adverse Events (participants affected / at risk) | 167/234 | 134/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=234) | Placebo (N=224)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine (N=234) | Placebo (N=224)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 8 (8) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (25) | 5 (5)
Dental caries (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (21) | 6 (6)
Saliva altered (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Calcinosis (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 2 (3) | 1 (1)
Malaise (General disorders) | 8 (9) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 14 (14) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 7 (7) | 2 (2)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 26 (33) | 39 (43)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Purulence (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (2)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 16 (18) | 7 (8)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 6 (6) | 3 (3)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Periarthritis calcarea (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Cartilage hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infrapatellar fat pad inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (9)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 15 (16) | 2 (2)
Dizziness postural (Nervous system disorders) | 4 (4) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 45 (45) | 16 (17)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep talking (Psychiatric disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/118 (1) | 0/121 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/116 (1) | 0/103 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/118 (1) | 1/121 (2)
Menstruation irregular (Reproductive system and breast disorders) | 0/118 (0) | 1/121 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days